CLINICAL TRIAL: NCT00890175
Title: Pulmonary Safety of Staccato® Loxapine for Inhalation in Subjects With Asthma
Brief Title: Staccato Loxapine Pulmonary Safety in Patients With Asthma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexza Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AMDC-004-105; 10 April 2009
Record Dates: First submitted 2009-04-27; First posted 2009-04-29 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2009-08

CONDITIONS: Asthma
Keywords: Asthma, Staccato loxapine
MeSH Terms: conditions — Asthma | interventions — Loxapine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Inhaled loxapine @ 0 & 10 h (Experimental): Inhalation of 10 mg of loxapine at 0 and 10 hours
  Interventions: Drug: Inhaled loxapine @ 0 & 10 h
- Inhaled placebo @ 2 & 10 hours (Placebo Comparator): Inhalation of 0 mg of loxapine (placebo) at 0 and 10 hours
  Interventions: Drug: Inhaled placebo @ 2 & 10 hours

INTERVENTIONS:
Drug: Inhaled loxapine @ 0 & 10 h — 10 mg, 2 doses, 10 hours apart
  Other Names: ADASUVE
  Arms: Inhaled loxapine @ 0 & 10 h
Drug: Inhaled placebo @ 2 & 10 hours — placebo, 2 doses, 10 hours apart
  Other Names: ADASUVE PLACEBO
  Arms: Inhaled placebo @ 2 & 10 hours

SUMMARY:
The purpose of this study is to assess the safety of 2 inhaled doses of Staccato Loxapine within a day in patients with asthma.

ELIGIBILITY:
Inclusion Criteria:

* History of mild to moderate persistent asthma for at least 6 months with pre-bronchodilator FEV1 ≥60% of predicted value.

Exclusion Criteria:

* History of COPD, or any other acute or chronic pulmonary disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2009-05; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Change in FEV1 from baseline by spirometry | at each post-treatment time point (15 min to 34 hr)

SECONDARY OUTCOMES:
Change in FVC from baseline by spirometry | at each post-treatment time point (15 min to 34 hr)
Treatment emergent adverse events | Post-treatment time points

CONTACTS AND LOCATIONS:
Overall Officials: Mildred D. Gottwald, PharmD, Study Director — Alexza Pharmaceuticals, Inc.
Locations (1):
- Allergy and Asthma Medical Group & Research Center, A.P.C., San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD submitted to regulatory authorities. Others may contact Alexza Pharmaceuticals, Inc. Please send your request to ClinicalTrialsInfo@alexza.com

REFERENCES:
- [Background] Gross N, Greos LS, Meltzer EO, Spangenthal S, Fishman RS, Spyker DA, Cassella JV. Safety and tolerability of inhaled loxapine in subjects with asthma and chronic obstructive pulmonary disease--two randomized controlled trials. J Aerosol Med Pulm Drug Deliv. 2014 Dec;27(6):478-87. doi: 10.1089/jamp.2013.1114. PMID 24745666